CLINICAL TRIAL: NCT03081013
Title: Randomized Controlled Trial of a Physical Activity Program for Teenagers (FIT-TEEN)
Brief Title: Randomized Controlled Trial of a Physical Activity Program for Teenagers
Acronym: FIT-TEEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Semra Ozdemir, Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSRNIG13nov007
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Physical Activity
Keywords: adolescents; social norms
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Private Arm (Active Comparator): At the end of each week, participants will be provided with the number of steps logged by the participants in their group. The number of steps will be ranked from highest to the lowest without any identifiable information about the participants.
  Interventions: Behavioral: Social information; Device: Fitbit
- Public Arm (Experimental): At the end of each week, participants will be provided with the number of steps logged by the participants in their group. The number of steps will be ranked from highest to the lowest with the full names of the participants corresponding to the number of steps.
  Interventions: Behavioral: Social information; Device: Fitbit

INTERVENTIONS:
Behavioral: Social information — Social comparison information will be provided to the study participants weekly via SMS
Device: Fitbit — Fitbit is a wireless pedometer that tracks steps of participants and will be offered in conjunction with a tailored website with customised information for participants.
  Other Names: Fitbit Flex, wireless pedometer, physical activity tracker

SUMMARY:
The study aims:

1. To test the effect of providing social comparison information on increasing physical activity among Singaporean adolescents.
2. To test whether providing social comparison information increases physical activity more when it is provided publicly compared to when it is provided anonymously.

DETAILED DESCRIPTION:
Childhood and adolescent obesity represents a major public health challenge worldwide. Singapore is no exception as the prevalence of obesity among children was estimated at 12%. Overweight and obese children are more likely to become obese adults, to develop non-communicable diseases at a younger age, and to have a shorter life expectancy. One of the main reasons behind the growing obesity epidemic is low levels of physical activity. Previous literature shows evidence of a steep decline in physical activity among boys after the primary school years and low levels of activity among girls throughout the primary and high school years in Singapore. Daily step counts are found to be up to 35% short of the recommended daily steps for adolescents. Low levels of physical activity are also associated with lower psychological well-being among adolescents. Thus, it is important that interventions aimed at increasing physical activity target adolescent years.

In this study, the investigators propose to test the effectiveness of providing social comparison information on increasing physical activity among adolescents. Participating adolescents will be randomized into a group and groups will be randomized into one of two study arms in a 4-month walking program:

Private arm: At the end of each week, participants will be provided with the number of steps logged by the participants in their group. The number of steps will be ranked from highest to the lowest without any identifiable information about the participants.

Public arm: At the end of each week, participants in this arm will be provided with the same information as in the other arm plus the names of the participants corresponding to the number of steps logged.

Social comparison information will be provided to the study participants via SMS. We will conduct a 4-month two-arm RCT to test whether social comparison information increases physical activity more when it is disclosed publicly compared to when it is provided anonymously. The primary outcome is the average number of steps taken per week by participants. Study outcomes relating to physical activity and health-related quality of life for participants will be evaluated at baseline and 4 months. Step activity will be tracked in real time via Fitbit wireless pedometers throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The study's target population is adolescents aged 13-16 years. Participants should be Singaporean citizens or permanent residents. Participants should be English-speaking. Participants should be willing to wear a pedometer for 4 months. Only participants who provide at least 8 (out of 14 days) valid days of pedometer data including at least 2 days of the weekend at baseline will be included.

Exclusion Criteria:

* Participants will be asked to complete a short screener questionnaire to ensure that they are healthy enough to participate. Participants reporting the following will be excluded:
* Having any medical condition that may limit their ability to walk as a means of physical activity
* Are unwilling to wear a wireless pedometer for 4 months

Participants will also be screened with a Physical Activity Readiness Questionnaire (PAR-Q). Those who answer 'YES' to any PAR-Q question will be permitted to enroll only if they provide written approval from a medical doctor.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The average number of steps taken per week by participants | 4 months
  These will be assessed through Fitbit pedometers at baseline and at the last 2 weeks of the trial. All participants will be issued a step counter, the Fitbit Flex™ for use during the entire 4-month RCT.

SECONDARY OUTCOMES:
Health Outcomes: Quality of life index | 4 months
  The quality of life will be assessed using the Pediatric Quality of Life Inventory (PedsQL) for adolescents. These measures will be taken twice; at baseline and at the end of the study.
Health Outcomes: Depression | 4 months
  Depression will be measured using Asian Adolescent Depression Scale (AADS) which is validated for Singaporean adolescents.These measures will be taken twice; at baseline and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Ozdemir, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Upon request from the principal investigator, individual participant data will be available to other researchers for secondary analysis purposes, such as meta-analyses, reanalysis or replication of results. Any data that will be shared will be de-identified so privacy of the participants will be protected.

REFERENCES:
- [Background] Must A, Strauss RS. Risks and consequences of childhood and adolescent obesity. Int J Obes Relat Metab Disord. 1999 Mar;23 Suppl 2:S2-11. doi: 10.1038/sj.ijo.0800852. PMID 10340798
- [Background] Chia M. Pedometer-assessed physical activity of Singaporean youths. Prev Med. 2010 May-Jun;50(5-6):262-4. doi: 10.1016/j.ypmed.2010.03.004. Epub 2010 Mar 11. PMID 20226810
- [Background] Lee KS, Trost SG. Validity and reliability of the 3-day physical activity recall in Singaporean adolescents. Res Q Exerc Sport. 2005 Mar;76(1):101-6. doi: 10.1080/02701367.2005.10599265. No abstract available. PMID 15810774
- [Background] Kirkcaldy BD, Shephard RJ, Siefen RG. The relationship between physical activity and self-image and problem behaviour among adolescents. Soc Psychiatry Psychiatr Epidemiol. 2002 Nov;37(11):544-50. doi: 10.1007/s00127-002-0554-7. PMID 12395145
- [Background] Sallis JF, Prochaska JJ, Taylor WC. A review of correlates of physical activity of children and adolescents. Med Sci Sports Exerc. 2000 May;32(5):963-75. doi: 10.1097/00005768-200005000-00014. PMID 10795788
- [Background] Maturo CC, Cunningham SA. Influence of friends on children's physical activity: a review. Am J Public Health. 2013 Jul;103(7):e23-38. doi: 10.2105/AJPH.2013.301366. Epub 2013 May 16. PMID 23678914
- [Background] Donaldson SI, Graham JW, Hansen WB. Testing the generalizability of intervening mechanism theories: understanding the effects of adolescent drug use prevention interventions. J Behav Med. 1994 Apr;17(2):195-216. doi: 10.1007/BF01858105. PMID 8035452
- [Background] Larimer ME, Neighbors C. Normative misperception and the impact of descriptive and injunctive norms on college student gambling. Psychol Addict Behav. 2003 Sep;17(3):235-43. doi: 10.1037/0893-164X.17.3.235. PMID 14498818
- [Background] Neighbors C, Larimer ME, Lewis MA. Targeting misperceptions of descriptive drinking norms: efficacy of a computer-delivered personalized normative feedback intervention. J Consult Clin Psychol. 2004 Jun;72(3):434-47. doi: 10.1037/0022-006X.72.3.434. PMID 15279527
- [Background] Schultz PW, Nolan JM, Cialdini RB, Goldstein NJ, Griskevicius V. The constructive, destructive, and reconstructive power of social norms. Psychol Sci. 2007 May;18(5):429-34. doi: 10.1111/j.1467-9280.2007.01917.x. PMID 17576283
- [Background] Yun D, Silk KJ. Social norms, self-identity, and attention to social comparison information in the context of exercise and healthy diet behavior. Health Commun. 2011 Apr;26(3):275-85. doi: 10.1080/10410236.2010.549814. PMID 21400325
- [Background] Tudor-Locke C, Craig CL, Beets MW, Belton S, Cardon GM, Duncan S, Hatano Y, Lubans DR, Olds TS, Raustorp A, Rowe DA, Spence JC, Tanaka S, Blair SN. How many steps/day are enough? for children and adolescents. Int J Behav Nutr Phys Act. 2011 Jul 28;8:78. doi: 10.1186/1479-5868-8-78. PMID 21798014
- [Background] Finkelstein EA, Tan YT, Malhotra R, Lee CF, Goh SS, Saw SM. A cluster randomized controlled trial of an incentive-based outdoor physical activity program. J Pediatr. 2013 Jul;163(1):167-72.e1. doi: 10.1016/j.jpeds.2013.01.009. Epub 2013 Feb 14. PMID 23415616
- [Background] Tudor-Locke C, Johnson WD, Katzmarzyk PT. Accelerometer-determined steps per day in US children and youth. Med Sci Sports Exerc. 2010 Dec;42(12):2244-50. doi: 10.1249/MSS.0b013e3181e32d7f. PMID 20421837
- [Background] Woo BS, Chang WC, Fung DS, Koh JB, Leong JS, Kee CH, Seah CK. Development and validation of a depression scale for Asian adolescents. J Adolesc. 2004 Dec;27(6):677-89. doi: 10.1016/j.adolescence.2003.12.004. PMID 15561310
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Saunders RP, Pate RR, Felton G, Dowda M, Weinrich MC, Ward DS, Parsons MA, Baranowski T. Development of questionnaires to measure psychosocial influences on children's physical activity. Prev Med. 1997 Mar-Apr;26(2):241-7. doi: 10.1006/pmed.1996.0134. PMID 9085394
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181
- [Derived] Lee JJ, Nadkarni NV, Teo I, Ozdemir S. The Effect of Social Norm-based Intervention with Observable Behaviour on Physical Activity among Adolescents: A Randomized Controlled Trial. BMC Sports Sci Med Rehabil. 2020 Aug 31;12:52. doi: 10.1186/s13102-020-00202-y. eCollection 2020. PMID 32874593
- See also: S'pore experts on the perils of childhood obesity and how to avert it." AsiaOne, 19 April 2014. — http://www.smu.edu.sg/sites/default/files/smu/news_room/smu_in_the_news/2014/sources/nov18/AsiaOne_20140419_1.pdf
- See also: Active for Life - Physical Activity: some is better than none." Health Promotion Board Singapore (HPB). — https://www.healthhub.sg/sites/assets/Assets/PDFs/HPB/PhysicalActivityPDFs/ActiveForLifebooklet_20110415_final.pdf